CLINICAL TRIAL: NCT06764303
Title: A Multicenter, Randomized, Open Label Phase II Clinical Trial Evaluating the Efficacy and Safety of NTQ5082 Capsules in the Treatment of Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: A Study of NTQ5082 Capsules in the Treatment of Paroxysmal Nocturnal Hemoglobinuria Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTQ5082-201
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 100mg qd (Experimental): This group included 12 subjects, all of whom received NTQ5082 capsules 100mg qd administration
  Interventions: Drug: NTQ5082 100mg qd
- 200mg qd (Experimental): This group included 12 subjects, all of whom received NTQ5082 capsules 200mg qd administration
  Interventions: Drug: NTQ5082 200mg qd

INTERVENTIONS:
Drug: NTQ5082 100mg qd — NTQ5082 100mg qd
  Arms: 100mg qd
Drug: NTQ5082 200mg qd — NTQ5082 200mg qd
  Arms: 200mg qd

SUMMARY:
NTQ5082 capsule is a small molecule CFB factor inhibitor. This study is a multicenter, randomized, open label phase II clinical trial aimed at evaluating the efficacy, safety, and PK/PD characteristics of NTQ5082 capsules in the treatment of patients with paroxysmal nocturnal hemoglobinuria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old (including lower limit), gender not limited.
2. According to the diagnostic criteria for PNH in the Chinese "Guidelines for the Diagnosis and Treatment of Rare Diseases" (2019 edition), subjects diagnosed with PNH have a red blood cell and/or granulocyte clone level of>10% within the 6 months prior to screening.
3. I have not received complement inhibitor treatment in the past.
4. Laboratory testing (local laboratory) shows that hemoglobin meets one of the following conditions: (1) screening period V1 and V2 (interval ≥ 7 days) hemoglobin<100g/L; (2) If the subject receives red blood cell transfusion treatment for PNH related anemia during the screening period, they must meet the condition of hemoglobin<100g/L at V1;
5. Screening periods V1 and V2 (with an interval of ≥ 7 days) were used to detect blood lactate dehydrogenase (LDH) levels (local laboratory)>1.5 times the upper limit of normal (ULN);
6. Vaccination with ACYW135 meningococcal and pneumococcal vaccines (if previously administered, effective titers should be provided) at least 14 days prior to the initial administration of the study drug (defined as D1); If vaccinated within 14 days before D1, prophylactic antibiotic treatment should be given until at least 14 days after vaccination;
7. Agree to use at least one effective contraceptive measure during sexual intercourse with their partner from the time of signing the informed consent form until 4 weeks after the last administration, and not to participate in sperm or egg donation.
8. Agree to sign the informed consent form and promise to comply with all regulations in the study.

Exclusion Criteria:

1. During the screening period, there was laboratory (local laboratory) evidence of bone marrow failure (reticulocyte count<100 × 109/L, platelet count<30 × 109/L, or neutrophil count<0.5 × 109/L).
2. During the screening period, the laboratory (local laboratory) results showed ALT or ALP>3 × ULN and the researcher deemed it unsuitable to participate in the study.
3. Prior to screening, the subject was receiving treatment with the following drugs, and the duration of treatment at the stable dose of the drug did not meet the following conditions: systemic use of corticosteroids for at least 4 weeks (≤ 15mg/day of prednisone or equivalent dose of corticosteroids); Iron supplements, vitamin B12, folic acid or androgens for at least 4 weeks; Vitamin K antagonists (such as warfarin) should be used for at least 4 weeks and the international normalized ratio (INR) should be stable; Low molecular weight heparin and oral anticoagulants (such as aspirin, rivaroxaban, idoxaban, apixaban) for at least 4 weeks; Erythropoietin (ESA), hypoxia inducible factor prolyl hydroxylase inhibitor (HIF-PHI), or immunosuppressant for at least 8 weeks.
4. Previous history of bone marrow/hematopoietic stem cell or solid organ transplantation (such as heart, lung, kidney, liver).
5. Individuals with a history of splenectomy or planning to undergo surgery during the trial period.
6. Previous history of meningococcal infection or active systemic bacterial, viral, or fungal infection within 14 days prior to the first administration of the study drug (defined as D1) (at the discretion of the investigator).
7. Patients with a history of malignant tumors within the past 5 years before screening, but those who have already been cured of local basal cell carcinoma of the skin, squamous cell carcinoma of the skin, papillary thyroid carcinoma, and cervical carcinoma in situ, are excluded.
8. Known or suspected genetic complement deficiency or primary or severe secondary immunodeficiency.
9. There is a history of clinically significant kidney, heart, liver, lung, and other conditions that the researchers have determined are not suitable for participation in this study, including but not limited to the following: severe uncontrolled hypertension, severe kidney disease (such as eGFR<30 mL/min/1.73m2), advanced heart disease (NYHA IV grade), severe lung disease (such as severe pulmonary arterial hypertension (WHO IV grade), unstable thrombotic events, etc.
10. Suffering from active hepatitis B (HBsAg positive and HBV-DNA>local laboratory detection limit), or hepatitis C (HCV antibody positive and HCV-RNA>local laboratory detection limit); Or tested positive for HIV; Or positive for Treponema pallidum antibody.
11. Have received any type of attenuated live vaccine within the previous 4 weeks of screening, or plan to receive any attenuated live vaccine during the research process.
12. Participated in any other interventional clinical trials (including drug and device clinical trials) within the previous 4 weeks prior to screening.
13. Suspect individuals who are allergic to the investigational drug or any of its components.
14. Pregnant and lactating female subjects.
15. Any medical condition that the researcher determines may affect the patient's participation in the study, may increase significant risks to the safety of the subjects, or other situations that the researcher determines are not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects whose hemoglobin (Hb) levels continue to increase by ≥ 20 g/L compared to baseline | 12 Weeks

SECONDARY OUTCOMES:
The proportion of subjects with Hb levels consistently ≥ 120 g/L | 12 Weeks
The proportion of subjects who did not receive blood transfusion | 12 Weeks
The number of red blood cell units transfused to the subjects receiving blood transfusion | 12 Weeks
Changes in Hb compared to baseline | 12 Weeks
Changes in reticulocyte count compared to baseline | 12 Weeks
Changes in lactate dehydrogenase (LDH) compared to baseline | 12 Weeks
Changes in total/indirect bilirubin compared to baseline | 12 Weeks
Changes in conjugated hemoglobin compared to baseline | 12 Weeks
Changes in free hemoglobin compared to baseline | 12 Weeks
The proportion of subjects with LDH<1.5 × ULN | 12 Weeks
Changes in Chronic Disease Treatment Functional Evaluation Fatigue (FACIT-F) Scale Score Compared to Baseline | 12 Weeks
Changes in the size of PNH red blood cell clones | 12 Weeks
Changes in the deposition of C3 complement protein fragments on PNH red blood cells | 12 Weeks
NTQ5082 capsule PD related biomarker levels: complement pathway activity, plasma fragment Bb, and human soluble terminal complement complex (sC5b-9) levels. | 12 Weeks
The Plasma concentration of NTQ5082 and metabolite NTQ5082-M in plasma under steady-state conditions (ss) | 12 Weeks
The incidence of breakthrough hemolysis in clinical practice. | 12 Weeks
The incidence of thromboembolic events. | 12 Weeks
Incidence and severity of adverse events | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: fengkui zhang, Principal Investigator — Hematology Hospital of the Chinese Academy of Medical Sciences; hongyan tong, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (2):
- China (2):
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang